CLINICAL TRIAL: NCT04330755
Title: The Effect of Levosimendan Versus Its Combination to Magnesium Sulphate on Spinal Cord Protection Guided by NIRS in Infants Undergoing Coarctectomy: A Randomized Controlled Study.
Brief Title: Levosimendan Versus Combination With Magnesium Sulphate on Spine Protection by NIRS in Infants Undergoing Coarctectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dalia Saad Abd-El Kader (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Dalia Saad Abd-El Kader, Principle investigator, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MD-223-2019
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2021-04

CONDITIONS: Aortic Coarctation
MeSH Terms: conditions — Aortic Coarctation | interventions — Saline Solution; Sodium Chloride; Simendan; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (Placebo Comparator): Control group will received saline
  Interventions: Drug: Saline Solution
- Group L (Active Comparator): Levosimendan group will received levosimendan infusion
  Interventions: Drug: Levosimendan
- Group M (Active Comparator): Levosimendan and Magnesium sulphate group will received both drugs
  Interventions: Drug: Levosimendan; Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Saline Solution — Placebo
  Other Names: Nacl 0.9 %
  Arms: Group C
Drug: Levosimendan — Levosimendan
  Arms: Group L; Group M
Drug: Magnesium Sulfate — Magnesium Sulfate
  Arms: Group M

SUMMARY:
In pediatric patients ,undergoing elective surgical correction of aortic coarcatation one of our main concern is spinal cord protection .Our aim to study the protective effect of levosimendan versus its combination with magnesium sulphate .

DETAILED DESCRIPTION:
Effect of levosimendan and its combination with magnesium sulphate infusion as spinal cord protection using NIRS values before Aortic cross clamp and 10,20 min after cross clamp till the end of surgery .

ELIGIBILITY:
Inclusion Criteria:

Age group ranging from 0 to 12 months of both sexes. Aortic coarcatation eligible for correction

Exclusion Criteria:

Parents or guardian refusal. Age more than12 months. Significant left ventricular dysfunction Patient with Heart block Patient with pre-existing CNS disorder eg seizure Patient with renal or hepatic dysfunction

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Near Infrared Spectroscopy value | Perioperative(immediately before cross clamp,10&20 min after cross clamping Aorta)
  After aortic cross clamping to compare the spinal cord protective effect of levosimendan versus its combination with magnesium sulphate.

CONTACTS AND LOCATIONS:
Overall Officials: Amel HY Abelala, professor, Study Chair — Cairo University
Locations (1):
- Sara ABD El-Salam, Cairo, Egypt